CLINICAL TRIAL: NCT00427466
Title: Multicenter Phase II Study With Pemetrexed in Patients With Pre-Treated Metastatic Soft Tissue Sarcomas
Brief Title: Pemetrexed in Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); German Sarcoma Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jth_006
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
The aims of this trial are to evaluate the efficacy and tolerability of pemetrexed in patients with metastatic soft tissue sarcoma who have progressed after or during an anthracycline-based chemotherapy and to assess the toxicity profile

DETAILED DESCRIPTION:
One therapy cycle takes a total of 3 weeks. On day 1, Pemetrexed is intravenously administered. The dosage is 500 mg/m2 over a period of 10 minutes. A repetition of this procedure is performed on day 22

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastasized or locally inoperable soft tissue sarcoma
* Progression or relapse after previous cytostatic treatment with adriamycin and/or an ifosfamide containing chemotherapeutic substance
* Two-dimensionally measurable/evaluable tumor parameters (according to WHO-criteria)
* Previous radiotherapy is acceptable as long as the irradiated area does not include the only measurable lesion
* Patient compliance and geographic proximity, which ensure the possibility of adequate Follow-up
* Life expectancy of more than 3 months
* ECOG <= 2
* Age at least 18 years
* Adequate bone marrow function at the initiation of therapy
* Adequate kidney function
* Patient consent
* Patient ability to consent

Exclusion Criteria:

* Previous or concurrent irradiation of the indicator lesion
* Other concomitant tumor therapy
* Severe impairment in hepatic function
* Active Infection
* Previous treatment with Pemetrexed
* Second tumor within the past 5 years (excepting basal cell carcinoma, adequately treated carcinoma in situ of the uterine cervix, of the bladder urothelium or colon polyps including pTis and pTin)
* Severely symptomatic cardiovascular and cerebrovascular disease
* HIV, active Hepatitis B or C
* Dementia, Cerebral stroke with cognitive deficits
* Kidney function <= 79 ml/min (calculated according to MDRD): Inability to interrupt treatment with NSAIDs/ASS/Cox-2 Inhibitors 2 days prior to and following administration of Pemetrexed. If a patient is taking an NSAID or salicylate with a long half-life it should not be taken five days prior to, on the day of or two days after application of Pemetrexed. Low dose acetyl salicylic acid administration is permitted (e.g. 100 mg/die.) There are no restrictions with kidney function greater than 80 ml/min.
* Inability or unwillingness to take folic acid, vitamin B12 or dexamethasone
* Pleural or pericardial exudate, ascites without a drain (3rd Space)
* Time Interval from the last course of chemotherapy < 4 weeks
* Symptomatic CNS-Metastases
* Gravidity or Lactation
* Women of reproductive age without reliable contraception if not the following applies: Must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen during and for 3 months after treatment
* Positive serum or urine pregnancy test
* Participation in another trial at the same time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Rate of response

SECONDARY OUTCOMES:
Rate of patients who are progression free at 3 and 6 months
Changes in median period of survival
Progression free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Joerg T Hartmann, MD, Principal Investigator — Medical Center II, University of Tuebingen, Germany
Locations (1):
- Medical Center II, University of Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Hartmann JT, Bauer S, Egerer G, Horger MS, Kopp HG, Grunwald V, Mayer F. Pemetrexed in patients with refractory soft tissue sarcoma: a non-comparative multicenter phase II study of the German Sarcoma Group AIO-STS 005. Invest New Drugs. 2013 Feb;31(1):167-74. doi: 10.1007/s10637-012-9840-8. Epub 2012 Jul 5. PMID 22763609